CLINICAL TRIAL: NCT03754283
Title: Transfer Accuracy of Indirectly Bonded Orthodontic Attachments With Vacuum Formed and Silicone Transfer Trays
Brief Title: Transfer Accuracy of Indirectly Bonded Orthodontic Braces With Different Transfer Trays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Dr. Cihan Aydoğan, Assistant prof, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-05.04.2016
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Malocclusion
Keywords: Indirect bonding; Accuracy
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone (Experimental): Indirect bonding performed with the silicone trays
  Interventions: Device: Indirect bonding
- Vacuum formed (Active Comparator): Indirect bonding performed with the vacuum formed trays
  Interventions: Device: Indirect bonding

INTERVENTIONS:
Device: Indirect bonding — Indirect bonding is the technique where orthodontic appliances are first placed on a model of the patient and then transferred to the patient using some kinf of trays

SUMMARY:
The aim of this study is to comparatively investigate the performances of two different and widely used transfer trays during indirect bonding of the orthodontic braces.

DETAILED DESCRIPTION:
The aim of the study is to compare the accuracy of orthodontic bracket and tube transfer between double layer silicone and double layer vacuum formed trays. The sample included 368 attachments bonded in 16 patients. Each patient received one silicone and one vacuum formed tray which were randomly allocated to provide 8 trays of each type for the upper and lower arches. 3D scan data and local best-fit alignments were used to calculate the translational and rotational movements of the orthodontic attachments. Chi-square and Mann-Whitney U tests were used to compare transfer accuracy and success between the groups.

ELIGIBILITY:
Inclusion Criteria:

* The presence of indication for both arches to be bonded in the same appointment

Exclusion Criteria:

* Presence of restorations, hypoplasia or decalcification on vestibular tooth surfaces
* Abnormal crown morphology

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Transfer accuracy (composite outcome) in milimetres and degrees. Which is measured on computer software. | Day 0 - Day 2
  The positional deviations between the attachments on the models and the mouth

CONTACTS AND LOCATIONS:
Locations (1):
- Cihan Aydoğan, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No